CLINICAL TRIAL: NCT01731210
Title: Clinical Evaluation Of The Nano Lv Lead System In Chronic Situation
Brief Title: Clinical Evaluation Of The Nano Lv Lead System In Chronic Situation (LENEA)
Acronym: LENEA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study stopped due to investigational device deficiency
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCNA02 - LENEA
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: LV Lead; LV Therapy; LV Treatment; LV Microcable

STUDY DESIGN:
Intervention Model Description: NANO LV lead
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: implantation of the new LV lead: NANO system.

SUMMARY:
The LENEA study is an international, prospective, open label, non-randomized multicenter clinical research study designed to assess the safety and effectiveness of the NANO LV lead system.

ELIGIBILITY:
Inclusion Criteria:

* Approved indication per ACC/AHA/HRS guidelines for implantation of a CRT-D system for treatment of heart failure or life threatening ventricular tachyarrhythmia(s)
* Receiving a new implant OR undergoing an upgrade from an existing ICD or pacemaker implant with no prior implanted LV lead OR undergoing a new LV implant attempt consecutive to a recent LV lead placement failure not related to coronary sinus cannulation failure
* Patient receiving the PARADYM RF CRT or PARADYM RF CRT SONR devices
* Ability to provide informed consent for study participation and is willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

* Ventricular tachyarrhythmia of transient or reversible causes such as acute myocardial infarction, digitalis intoxication, drowning, electrocution, electrolyte imbalance, hypoxia or sepsis, uncorrected at the time of the enrolment;
* Incessant Ventricular tachyarrhythmias;
* Unstable angina, or acute MI , CABG , or PTCA within the past 4 weeks;
* Correctable valvular disease that is the primary cause of heart failure;
* Post heart transplant (patients who are waiting for a heart transplant are allowed in the study);
* Patient who had previously a permanently implanted LV lead;
* Concurrent implant with another pacemaker or ICD (previously implanted pacemaker or ICD devices should be removed prior to implant with the Paradym RF CRT-D or Paradym RF CRT SONR);
* Already included in another clinical study that could confound the results of this study;
* Life expectancy less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-10-31 (Actual); Study Completion 2013-12-19 (Actual)

PRIMARY OUTCOMES:
Freedom from left ventricular lead related complications through 1 month | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Charles Nicolle, Rouen, France